CLINICAL TRIAL: NCT06057454
Title: Evaluating the Safety and Tolerability of R-5280 in Mitigating Type 1 Diabetes in Newly Diagnosed Patients
Brief Title: R-5280 in Newly Diagnosed Patients With Type 1 Diabetes
Acronym: R-5280
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rise Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RISE R-5280
Record Dates: First submitted 2023-09-15; First posted 2023-09-28 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes; Type 1 Diabetes (Juvenile Onset); Diabetes Mellitus, Type 1
Keywords: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Double Blinided, placebo controlled, Phase 1B study.
Who Masked: Participant, Investigator
Masking Description: Double blind placebo controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator): R-5280, Taken Twice a day, orally with food for 12 weeks (84 days)
  Interventions: Drug: R-5280
- Placebo Comparator (Placebo Comparator): Food starch, taken twice a day, orally with food for 12 weeks (84 days)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: R-5280 — Modified Superior Starch
  Arms: Active Comparator
Other: Placebo — Food Grade Starch
  Arms: Placebo Comparator

SUMMARY:
Evaluating the adverse events and tolerance of R-5280 in Mitigating Type 1 Diabetes in Newly Diagnosed Patients

DETAILED DESCRIPTION:
Double blinded, placebo controlled, Phase 1B study assessing the safety and efficacy of 12 weeks daily administrations of R-5280 in newly diagnosed Type 1 Diabetes adolescents

ELIGIBILITY:
Inclusion Criteria:

* Newly Diagnosed children (age 11-17 years old)
* BMI <85%
* Diagnosed by ADA criteria with T1D within 2 years
* Accepted to adhere to a healthy diabetic diet as recommended by the ADA

Exclusion Criteria:

* Monogenic forms of diabetes or type 2 diabetes
* History of ongoing infection or antibiotic treatment within the past four (4) weeks
* History of immunocompromised, recurrent infections, steroid intake (inhaled or oral forms) or other immunosuppressant use in the past six (6) months
* History of chronic gastrointestinal disease, possible or confirmed celiac disease
* Pregnancy or possible pregnancy
* Allergy to corn (prebiotic), milk allergy, soy (present in the MMTT meal) or their products
* Participation in other intervention research trials within the past three (3) months
* Anticipated major change in diabetes management during the study (e.g., change from injections to insulin pump therapy or new continuous monitor usage, all known to significantly alter glycemia)
* Children consuming a high-fiber or vegetarian diet (consuming three (3) or more servings of high fiber foods on four (4) or more days per week) or any fiber supplements will be excluded (to be assessed at screening)
* Any COVID vaccines within 30 days prior to Day 1

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Measurement of adverse events from the date of the first dose through 12 weeks of R-5280 tolerance | 12 Weeks
  The number of participants with treatment-related adverse events as evaluated by CTCAE v5.0, will be reviewed to see the results from baseline in toxicology scores at 12 Weeks compared to placebo.

SECONDARY OUTCOMES:
Measurement of clinical activity and to determine the gut microbiome profile in youth with recently diagnosed Type 1 Diabetes | 12 Weeks
  To measure the levels of glucose (in milligrams) in the blood at the beginning and again at 12 weeks, and the measurement of C-Peptide (in nanograms) in the blood at the beginning and again at 12 weeks versus placebo, changes in the type of gut bacteria at the beginning and again at 12 weeks versus placebo.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Edward Jenner Research Group LLC, Plantation, Florida
  - Mayo Clinic, Rochester, Minnesota
  - UTSW Medical Center, Dallas, Texas